CLINICAL TRIAL: NCT02385552
Title: Seoul National University Hospital Healthcare System Gangnam Center Colonoscopy Quality Upgrade Project (Gangnam-CUP): Development of Quality Indicators and Quality Improvement Plan of Colonoscopy in Experienced Endoscopist.
Brief Title: Development of Quality Indicators and Quality Improvement Plan of Colonoscopy in Experienced Endoscopist
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Associate Professor, Seoul National University Hospital
Other Study IDs: H-1502-003-644
Record Dates: First submitted 2015-03-01; First posted 2015-03-11 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Colonic Polyps; Colonic Neoplasms
Keywords: colonoscopy; quality improvement; adenoma detection rate
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Experienced endoscopists: All of the experienced endoscopists will receive feedbacks from investigators about their own adenoma detection rate every 3 months
  Interventions: Behavioral: Feedback

INTERVENTIONS:
Behavioral: Feedback — Experienced endoscopists will receive feedbacks from investigators about their own adenoma detection rates.

SUMMARY:
The purpose of this study is to determine clinical factors affecting quality indicators of colonoscopy including adenoma detection rate, and whether quality of colonoscopy could be elevated by improving related factors.

DETAILED DESCRIPTION:
This study is an extension of quality assurance program in Seoul National University Hospital Healthcare System Gangnam Center. This study is composed of five periods. First, quality indicators of colonoscopy in experienced endoscopists will be analyzed retrospectively from January 2011 to december 2014. Individual differences and changes of quality indicators in every endoscopist will be verified. In second period, from January 2015 to March 2015, quality assurance program will be activated. Endoscopists will be educated by EQUIP (Endoscopic Quality Improvement Program). Also split-regimen bowel preparation instead of same-day regimen and Boston bowel preparation scale will be introduced to standardize disparity of grading. Third, prospective trial starts from April 2015 to March 2018. All endoscopists will receive feedbacks of their own adenoma detection rates in every 3 months. Changes of quality indicators for each endoscopist will be investigated, and annually monitored by institutional review board. If there is a significant improvement of quality indicators in interim assessment, prospective trial will be extended until April 2018. Fourth is wash-out period from April 2018 to march 2019. Feedbacks will be stopped and adenoma detection rates and quality indicators of endoscopists will be compared with those from prospective period. Finally, cumulative rate and mortality rate of colorectal cancers will be investigated until December 2019.

ELIGIBILITY:
Inclusion Criteria:

* Customers who received colonoscopy in Seoul National University Hospital Healthcare System Gangnam Center from 2011 to 2019.

Exclusion Criteria:

* Age <18 years
* Customers who refused to offer their health check up data
* History of inflammatory bowel disease
* History of familial adenomatous polyposis
* Customers who received Incomplete colonoscopy
* History of previous colorectal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Customers who received colonoscopy in Seoul National University Hospital Healthcare System Gangnam Center from 2011 to 2019.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2011-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 8 years
  (total, right, transverse, left)

SECONDARY OUTCOMES:
Colonoscopy performance indicators | 8 years
  Colonoscopy withdrawal time in negative complete colonoscopy
Colonoscopy performance indicators | 8 years
  The number of taken pictures in negative complete colonoscopy
Colonoscopy performance indicators | 8 years
  The position changes during colonoscope insertion and withdrawal
Colonoscopy quality indicators | 8 years
  Colorectal cancer detection rate
Colonoscopy quality indicators | 8 years
  Advanced adenoma detection rate
Colonoscopy quality indicators | 8 years
  Adenoma detection rate plus
Colonoscopy quality indicators | 8 years
  Polyp detection rate (total, right, transverse, left)
Colonoscopy quality indicators | 8 years
  Multiple adenoma detection rate
Colonoscopy quality indicators | 8 years
  Serrated polyp detection rate (total, right, transverse, left)
Colonoscopy quality indicators | 8 years
  Complication rate (bleeding, perforation, pain)

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Chung, M.D., Ph.D., Principal Investigator — Department of Internal Medicine and Healthcare Research Institute, Healthcare System Gangnam Center, Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Healthcare System Gangnam Center, Seoul National University Hospital, Seoul
  - Ji Yeon Seo, Seoul